CLINICAL TRIAL: NCT05305469
Title: Early Identification and Prognosis Prediction of Sepsis Through Multiomics
Acronym: EIPPSM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yantai Yuhuangding Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-031
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Sepsis
Keywords: Prognosis; Inflammation; Immune; Multiomics; Machine learning
MeSH Terms: conditions — Sepsis; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine, and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- GN: Gram-negative bacteria infection group
- GP: Gram-positive bacteria infection group
- Fungal: Fungal infection group
- Viral: Viral infection group
- Control: Non-sepsis group

SUMMARY:
This study aims to integrate multi-omics data and clinical indicators to reveal pathogen-specific molecular patterns in patients with sepsis and establish prognostic prediction models through multiple machine learning algorithms.

DETAILED DESCRIPTION:
This study aims to quantify the plasma metabolome, single nucleotide polymorphisms (SNPs) of exons and immunocytokines of septic patients with different pathogen infections and prognostic outcomes. Multi-omics data, cytokines, and clinical indicators will be integrated through multiple machine learning algorithms to reveal pathogen-specific molecular patterns and multi-dimensional prognostic prediction models.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sepsis or septic shock who meet the diagnostic criteria (2016 sepsis 3.0 standard);
* Age 18～85 years old.

Exclusion Criteria:

* ICU stay of the subjects less than 72 hours;
* Female subjects who are pregnant;
* The subjects not sure if infected;
* The subjects performed CPR;
* The subjects suffer from chronic renal disease;
* The subjects with incomplete clinical data.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study cases are from the Department of Critical Care Medicine, a top-grade hospital in Yantai
Sampling Method: Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathogen-specific patterns | March 2022 - December 2023
  To elucidate the unique infection pathogen-specific molecular patterns in septic patients

SECONDARY OUTCOMES:
Prognostic prediction models | March 2022 - December 2024
  To establish the models using multi-omics data to predict the prognosis of sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Jing Wang, Principal Investigator — Yantai Yuhuangding Hospital
Locations (1):
- Yantai Yuhuangding Hospital, Yantai, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang J, Sun Y, Teng S, Li K. Prediction of sepsis mortality using metabolite biomarkers in the blood: a meta-analysis of death-related pathways and prospective validation. BMC Med. 2020 Apr 15;18(1):83. doi: 10.1186/s12916-020-01546-5. PMID 32290837